CLINICAL TRIAL: NCT03710031
Title: Developing the Bio-behavioral Foundation for Self-Management of Psycho-neurological Symptoms in Hematopoietic Cell Transplant (HCT) Survivors
Brief Title: Developing Self-Management Interventions After HCT
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201802329; R21NR017749 (NIH); OCR18772 (Other: University of Florida)
Record Dates: First submitted 2018-09-26; First posted 2018-10-17 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Hematopoietic Stem Cell Transplant (HSCT)
Keywords: psychoneurological symptoms (PNS); quality of life (QOL); hematopoietic stem cell transplant (HSCT); microbiota gut-brain axis; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiome: Stool, Cytokines and C-Reactive Protein: Blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSCT Survivors: PNS tracking will occur through blood and stool samples to track the interplay among psychoneurologic symptoms (PNS) as they relate to diminished QOL among survivors of HSCT.
  Interventions: Other: PNS Tracking

INTERVENTIONS:
Other: PNS Tracking — Through blood and stool samples the study team will track the interplay among PNS as they relate to diminished QOL. Symptoms tracked include neurocognitive dysfunction, fatigue, anxiety, depression and pain, inflammation (cytokines and C-reactive protein), gut microbiota [(GM) richness and diversity] and diet (macronutrients: carbohydrates, fats and proteins).

SUMMARY:
This is a prospective, longitudinal, observational trial to evaluate quality of life in hematopoietic stem cell transplant survivors.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplant (HSCT) survival rates continue to increase as treatment protocols improve. However, HSCT survivors face many mental, emotional, and physical challenges that threaten quality of life (QOL), which, according to the American Society of Clinical Oncology, is the most important treatment outcome next to survival. Psychoneurologic symptoms (PNS) significantly diminish QOL after HSCT. PNS often co-occur and may be associated with inflammation related to perturbations of the gut microbiota. This project will track the interplay among these factors in 50 adult survivors of HSCT to lay the groundwork for a targeted dietary self-management intervention to mitigate PN symptoms.This is to be achieved by elucidating the complex bio-behavioral mechanisms of distressing symptoms in HCT patients such as neurocognitive dysfunction, fatigue, anxiety, depression and pain, inflammation (cytokines and C-reactive protein), gut microbiota [(GM) richness and diversity] and diet (macronutrients: carbohydrates, fats and proteins).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for HSCT with the Bone Marrow Transplant Program at the UF Health Cancer Center (UFHCC) [specifically bone marrow diseases, myelodysplastic-myeloproliferative diseases, lymphoma, bone marrow neoplasm or leukemia]
* Written informed consent obtained from the subject to take Mini-Mental State Examination (MMSE) prior to enrollment on the study and to comply with all the study-related procedures.
* Score at least a 24 on the Mini-Mental State Examination (MMSE) prior to enrollment

Exclusion Criteria:

* Subjects with any of the following will not be eligible for study participation:
* Patient has prior history of HSCT
* Patient has diagnosis that could interfere with neurocognitive function such as dementia, a concurrent diagnosis of systemic lupus erythematous or multiple sclerosis, diagnosis of a major depressive disorder, schizophrenia or untreated bipolar disease.
* Pregnant women are not eligible for transplant therefore will not be enrolled on the study
* Inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematopoietic Stem Cell Transplant (HSCT) Survivors. Survival rates continue to increase as treatment protocols improve; by 2030, an estimated half-million HSCT recipients in the United States will be long-term survivors. However, HSCT survivors continue to face many mental, emotional, and physical challenges that threaten QOL, which, according to the American Society of Clinical Oncology, is the most important treatment outcome next to survival. Therefore, a prospective, observational design to longitudinally examine these factors in 50 adult (at least 18 years of age) survivors of HSCT to lay the groundwork for the future development of a targeted dietary self-management intervention to mitigate PN symptoms in this growing group of HSCT survivors is being planned.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels of inflammatory markers (cytokines and CRP) of individuals post allogeneic HSCT | Baseline; Day 30; Day 100
  Cytokines will be analyzed using a multiplex assay by Millipore Company. Compared to the traditional enzyme-linked immunosorbant assays (ELISA), the multiplex is comparable and more sensitive to lower concentration levels of cytokines than the ELISA. One laser identifies a specific bead and another laser identifies the reported antibody associated with the bead-bound cytokine. One hundred beads for each of the 17 cytokines in every sample are assayed and a mean cytokine binding for the sample is determined. The manufacturer reports that the assay accurately measures cytokine values in a range of 1-2500pg/ml. Serum CRP will be measured using the ALPCO's (American Laboratory Products Company) high-sensitivity CRP assay which uses latex particle enhanced immunoturbidimetry for quantitative CRP determination.
Change in diversity and levels of fecal microbes of individuals post allogeneic HSCT | Baseline; Day 30; Day 100
  Fecal microbial DNA will be extracted from between 50-200 mg of fecal material. The 16S ribosomal gene (V4 region) of each sample will be amplified using a barcoding system to allow multiplexing with the Illumina MiSeq system. We will use UNIFRAC algorithm to evaluate the null hypothesis that the structure of the microbial community is insensitive to cGVHD and symptoms of cGVHD. Differences in taxa are implicated by our high throughput sequencing methods will be confirmed by other techniques including culturing (where appropriate) and qPCR with taxa-specific primers.
Change in behavioral responses (symptoms) of individuals post allogeneic HSCT | Baseline; Day 30; Day 100

SECONDARY OUTCOMES:
Health Promoting Lifestyle Profile II (HPLPII) | Baseline; Day 30; Day 100
  The Health Promoting Lifestyle Profile II (HPLPII) will be used to identify lifestyle choices that may affect relationships and differences between groups. HPLPII measures health promoting behaviors across several dimensions with subscales of health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations and stress management. This is a 52-item summated behavior rating scale using a 4-point response format to measure the frequency of self-reported health-promoting behaviors. It is a well validated toll and takes approximately 10 minutes to complete.
Brief Pain Inventory (BPI) | Baseline; Day 30; Day 100
  Pain will be assessed using the Brief Pain Inventory (BPI). The BPI was created to evaluate two dimensions of pain: 1) the severity and 2) the interference. This tool is well validated with Cronbach's alpha .80-.87 pain severity and .89-.92 for interference.22 The BPI consists of a body diagram to indicate location of pain and a general question asking if pain is present. Four items assess pain intensity or severity and seven item s assess pain interference. Both use an eleven point scale ranging from 0 (no pain or interference) to 10 (worst pain or interference). This instrument takes approximate five minutes to complete.
Hospital Anxiety and Depression Scale (HADS) | Baseline; Day 30; Day 100
  Depressive symptoms will be assessed using the subscale for depression from the Hospital Anxiety and Depression Scale (HADS). 23This instrument is used to assess the presence and severity of anxiety and depressive symptoms over a seven day period. The depression subscale is comprised of seven items using a four point scale ranging from 0 (least severe) to 3 (most severe). Cronbach's alpha has been found to be high (.82-.90) for the HADS depression subscale.
Brief Fatigue Inventory (BFI) | Baseline; Day 30; Day 100
  Fatigue will be assessed using the Brief Fatigue Inventory (BFI). The BFI is a nine item, eleven point scale that assesses physical, affective, cognitive and social domains in a two dimensions, fatigue intensity and interference. Severity scores are as follows: 1) mild (1-3), 2) moderate (4-6) and 3) severe (7-10). This tool is well establish and validated. The Cronbach's alpha ranged from .95-.96 for individual items and an internal consistency of .96 overall. The questionnaire takes approximately five minutes to complete and a global score can be ascertained by averaging the total score.
Memorial Symptom Assessment Scale (MSAS-SF) | Baseline; Day 30; Day 100
  To comprehensively explore symptoms, the Memorial Symptom Assessment Scale (MSAS-SF) will be used to measure multiple dimensions (frequency, severity, and distress) of 32 common cancer symptoms. The Cronbach alpha for the MSAS-SF subscales ranged from .76-.86 and the test-retest correlation coefficients ranged from .86-.94 at one day and one week respectively. The total time to complete this form is approximately 10 minutes. This form allows for patients to identify and quantify "other" symptoms.
Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) | Baseline; Day 30; Day 100
  Health related quality of life (HRQOL) will be measured using the Functional Assessment of Cancer Therapy- Bone Marrow Transplantation (FACT-BMT). This is a well validated HRQOL measure. This is a 27-item questionnaire asking questions across four domains: physical well-being, social well-being, emotional well-being and functional well-being. This measure takes about 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Kelly, PhD, RN, OCN, Principal Investigator — College of Nursing, University of Florida
Locations (1):
- UF Health Cancer Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kelly DL, Lyon DE, Yoon SL, Horgas AL. The Microbiome and Cancer: Implications for Oncology Nursing Science. Cancer Nurs. 2016 May-Jun;39(3):E56-62. doi: 10.1097/NCC.0000000000000286. PMID 26110573